CLINICAL TRIAL: NCT04743453
Title: EFFECT OF ADDING DAPAGLIFLOZIN TO ALLOGRAFT DYSFUNCTION OF RENAL TRANSPLANTED PATIENTS: A Prospective, Randomized, Single-blinded, Placebo- Controlled Study.
Brief Title: EFFECT OF ADDING DAPAGLIFLOZIN TO ALLOGRAFT DYSFUNCTION OF RENAL TRANSPLANTED PATIENTS.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41012620.6.1001.0068
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Kidney Transplantation; Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Kidney Transplantation; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to add either Dapagliflozin 10 mg or Placebo to their treatment. Study drug will be administered by once-daily orallly.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg: Study drug will be administered by once-daily orallly. The first dose MUST be started within 1 and 7 days after randomization. The subsequent doses will be administered 24 ± 4 hours after the previous dose.
  Arms: Dapagliflozin
Drug: Placebo — Placebo will be administered by once-daily orallly. The first dose MUST be started within 1 and 7 days after randomization. The subsequent doses will be administered 24 ± 4 hours after the previous dose.
  Arms: Placebo

SUMMARY:
Sodium-glucose co-transporter 2 (SGLT2) inhibitors reduce plasma glucose and haemoglobin A1c(HbA1c) in patients with type 2 diabetes mellitus by increasing urinary glucose excretion in a non-insulin-dependent fashion.

However, in some situations lead to a diminished number of functional glomeruli with a consequent hyperfiltration in the remaining ones. This fact may be where the use of SGLT2 inhibitor could attenuate the renal damage.

The purpose of our study is to evaluate the impact of using dapagliflozin on the renal functional deterioration of renal transplanted patients diabetics or not.

This is a prospective, randomized, single-blinded, double-center, controlled trial.

Patients will be randomized to add either Dapagliflozin 10 mg or Placebo to their treatment. Study drug will be administered by once-daily orallly. The first dose MUST be started within 1 and 7 days after randomization. The subsequent doses will be administered 24 ± 4 hours after the previous dose.

ELIGIBILITY:
Inclusion Criteria:

1. Renal Transplanted patients with one to 5 years after transplantation, being followed at the out-patient clinics of the HCFMUSP and HRim;
2. ≥18years of age;
3. 45 ≥ eGFR ≥ 25 mL/min/1.73m2 or 45<eGFR<60 ml/min/1.73m2 with a loss of eGFR of ≥10% in the last year.

Exclusion Criteria:

1. Type 1 diabetes;
2. New York Heart Association Class IV congestive heart failure;
3. Myocardial infarction, unstable angina, stroke or transient ischaemic attack within 8 weeks prior to enrolment;
4. Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or valvular repair/replacement within 8weeks prior to enrolment;
5. Any condition outside the renal and cardiovascular study area with a life expectancy of < 1 year based on investigator's clinical judgement;
6. Hepatic impairment [aspartate transaminase or alanine transaminase >3 times the upper limit of normal (ULN) or total bilirubin >2 times the ULN at the time of enrolment;
7. Acute or chronic antibody mediated rejection;
8. Albuminuria due to other causes (mTOR inhibitors, Polyoma nephropathy, lymphoproliferative disorder etc…)
9. Patients with a previous medical history of recurrent urinary tract infections or severe genital infection;
10. Renal biopsies showing acute or chronic anti-body mediated rejection, transplant glomerulopathy, BKV nephropathy.
11. Patients under any other IS regimen besides Tacrolimus/MPA/Steroids
12. Pregnant patients as well as those breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the mean ΔmGFR, between baseline and one year after randomization. | 12 months
  To evaluate the mean ΔmGFR, between baseline and one year after randomization between groups: Dapaglifozin and Placebo groups. (ΔmGFR is defind as the difference between measured GFR (mGFR) at baseline and at one year).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas - FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill M, Leung M, Luo CY, Cheung C, Beauchesne A, Chang D, Lan J, Johnston O. Erythrocytosis and thrombotic events in kidney transplant recipients prescribed a sodium glucose cotransport-2 inhibitor. Clin Transplant. 2023 Aug;37(8):e15013. doi: 10.1111/ctr.15013. Epub 2023 May 11. PMID 37170711